CLINICAL TRIAL: NCT06852287
Title: Phase II Clinical Study of GemOX Hepatic Arterial Infusion Combined with Lenvatinib and Toripalimab for Advanced and Unresectable Intrahepatic Cholangiocarcinoma and Gallbladder Cancer
Acronym: GOLD-HAIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Wei Zhang, Surgical chief physician & Deputy Director of Hepatobiliary Oncology Department, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20241047; GOLD-HAIC (Other: Tianjin Medical University Cancer Institute and Hospital)
Record Dates: First submitted 2024-10-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Intrahepatic Cholangiocarcinoma (Icc); Gall Bladder Cancer
Keywords: GemOX, Lenvatinib, Toripalimab
MeSH Terms: conditions — Cholangiocarcinoma; Cirrhosis, Familial, with Pulmonary Hypertension; Gallbladder Neoplasms | interventions — Drug Therapy; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GemOX hepatic arterial infusion combined with lenvatinib and Toripalimab (Experimental): Triprolizumab: 240mg ivd d1, q3w; Lenvatinib: 8-12mg po qd (body weight<60kg, 8mg po qd; body weight ≥ 60kg, 12mg po qd); Chemotherapy hepatic arterial infusion (GOLD HAIC): d1 oxaliplatin: 100-125mg+gemcitabine: 800-1000mg; q3w.
  Interventions: Drug: chemotherapy with gemcitabine and oxaliplatin; small molecure TKI lenvatinib; immune-checkpoint inhibitor toripalimab.

INTERVENTIONS:
Drug: chemotherapy with gemcitabine and oxaliplatin; small molecure TKI lenvatinib; immune-checkpoint inhibitor toripalimab. — Toripalimab: 240mg ivd d1, q3w; Lenvatinib: 8-12mg po qd (body weight<60kg, 8mg po qd; body weight ≥ 60kg, 12mg po qd) Chemotherapy by hepatic arterial infusion (GOLD HAIC): d1 oxaliplatin: 100-125mg+gemcitabine: 800-1000mg; q3w.

SUMMARY:
For advanced unresectable intrahepatic cholangiocarcinoma and gallbladder cancer, the current standard first-line treatment is a combination of chemotherapy and immunotherapy. However, the efficacy rates remain low. Hepatic artery infusion chemotherapy can reduce systemic drug dosages while increasing local drug concentrations, which is expected to enhance overall efficacy and minimize drug toxicity and side effects.

This study utilized a hepatic artery infusion chemotherapy regimen that combines gemcitabine with oxaliplatin, along with the small molecule tyrosine kinase inhibitor lenvatinib and the immune checkpoint inhibitor toripalimab. The aim was to improve treatment efficacy and create opportunities for conversion surgery. The primary endpoint was the objective response rate, while the secondary endpoints included the surgical resection rate, complete pathological response rate (pCR), overall survival (OS), and the incidence of adverse reactions.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 or above
2. Histopathological or cytological diagnosis of intrahepatic cholangiocarcinoma or gallbladder cancer
3. A tumor that cannot be removed by three independent surgeons.
4. Expected lifespan ≥ 12 weeks
5. ECOG PS score 0-1 points
6. The patient voluntarily participates and signs an informed consent form;
7. Expected compliance is good, able to follow up on efficacy and adverse reactions according to the protocol requirements.

Exclusion criteria:

1. Use any systemic research anti-cancer drugs
2. Active autoimmune diseases or a history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (which may include hormone replacement therapy)
3. Asthma requires the use of bronchodilators for medical intervention
4. Congenital or acquired immune dysfunction, such as human immunodeficiency virus (HIV) infection
5. Clinical symptoms or uncontrolled heart disease
6. Severe infection within 4 weeks before the first use of medication
7. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
8. Vaccination with attenuated live vaccine within 4 weeks before treatment
9. Other systemic malignant tumors in the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | through study completion, an average of 1 year
  Objective Response Rate (ORR) is a key metric commonly used to assess the efficacy of cancer treatments, especially in clinical trials. It primarily measures the proportion of patients who exhibit a significant reduction in tumor size following treatment. Here's a detailed explanation of ORR:
  1. Definition: ORR refers to the percentage of patients who experience a notable reduction in tumor size within a specified timeframe after receiving treatment. It typically encompasses two types of responses:
     Complete Response (CR): The tumor completely disappears, confirmed by follow-up assessments showing no measurable tumor.
     Partial Response (PR): The tumor size is reduced by a certain percentage (usually 30% or more), but measurable tumor remains.
  2. Calculation Method
  The formula for calculating ORR is as follows:
  ORR=CR+PR.

SECONDARY OUTCOMES:
Surgical resection rate | through study completion, an average of 1 year
  Surgical resection rate is the proportion of patients who underwent surgical resection among all patients
Pathological complete response rate (pCR rate) | through study completion, an average of 1 year
  Pathological complete response rate (pCR rate) is the proportion of patients who underwent surgical resection who achieved pathological complete response.
Overall survival (OS) | through study completion, an average of 5 years
  Overall survival time (OS) is the time from enrollment in clinical trials to patient death or loss to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tia, China

IPD SHARING:
Plan to Share IPD: No